CLINICAL TRIAL: NCT06460883
Title: Effects of Eccentric Banded Leg Curls Versus Eccentric Cable Leg Curls Exercises on Eccentric Knee-flexor Strength, Power and Endurance in Cricket Players
Brief Title: Effects of Eccentric Banded Leg Curls Versus Eccentric Cable Leg Curls Exercises in Cricket Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/01103
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Hamstring Muscle; Muscle Strength; Treatment Efficacy
Keywords: Eccentric hamstring device; Hamstring strain; Lengthened state eccentrics; Nordbord; Eccentric banded leg curls; Eccentric cable leg curls

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eccentric cable leg curls (Experimental): Group A players will perform eccentric cable leg curls
  Interventions: Other: eccentric cable leg curls
- eccentric banded leg curls (Active Comparator): Group A players will perform eccentric banded leg curls
  Interventions: Other: eccentric banded leg curls

INTERVENTIONS:
Other: eccentric cable leg curls — The players will undergo eccentric cable leg curls, completing 15 reps of 3 sets every other day with 30-45 seconds rest between sets, a total duration of 40 minutes conducted four days a week over a four-month training period.
  Arms: eccentric cable leg curls
Other: eccentric banded leg curls — The players will undergo eccentric banded leg curls, completing 15 reps of 3 sets every other day with 30-45 seconds rest between sets, a total duration of 40 minutes conducted four days a week over a four-month training period.
  Arms: eccentric banded leg curls

SUMMARY:
Hamstring injuries are highly prevalent among cricket players, comprising 10% of all injuries in field-based team sports. Eccentric strength deficits and imbalances in muscle strength are linked to a higher risk of such injuries. Our randomized clinical trial aims to assess eccentric hamstring strength using eccentric banded leg curls and eccentric cable leg curl exercises, measured by the Nordbord device. This tool provides accurate measurements of eccentric hamstring strength, power, and endurance, crucial for injury prevention in athletes. Thirty-two male professional cricketers will participate, divided into two groups receiving different exercise plans. Each group will perform 15 reps in 3 sets with rest intervals, four times a week for four months. The Nordbord device will assess hamstring strength before and after the exercise plan. Statistical analysis will be done using SPSS V25, employing descriptive statistics for frequency distribution and inferential statistics such as t-tests to compare outcomes between treatment groups.

DETAILED DESCRIPTION:
The present study aims to assess the effects of eccentric banded leg curls versus eccentric cable leg curls exercise on eccentric knee-flexor strength assessed with an instrumented Nordic hamstring device (Nordbord) after training in Cricket Players.

ELIGIBILITY:
Inclusion Criteria:

* Participants range in age from 14 to 35 years.
* Only male individuals are eligible for inclusion.
* Eligible participants include professional cricketers at domestic and international levels (U-16, U-19, or above), as well as recent additions to domestic cricket.
* Participants must have either good health or chronic lower extremity injuries impacting hamstring muscle strength.
* Willingness to provide informed consent is a prerequisite for study participation.

Exclusion Criteria:

* Individuals outside the age range of 14 to 35 years are excluded.
* Exclusion criteria include a medical history of neurological or musculoskeletal conditions impacting the lower extremities, such as nerve disorders or severe arthritis.
* Those with lower extremity injuries sustained within the previous two months are ineligible.
* Participants who have undergone lower extremity surgery within the past six months are not eligible.
* Exclusion applies to individuals taking medications that may impact muscle strength or neuromuscular function.
* Individuals who refuse to provide informed consent are not included in the study.

Ages: 14 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2024-12-18 (Actual); Primary Completion 2025-04-05 (Actual); Study Completion 2025-04-09 (Actual)

PRIMARY OUTCOMES:
Eccentric hamstring strength | 4 months
  The NordBord is a great tool for measuring hamstring strength of each leg allowing for tracking of overall strength gains and side-to-side imbalances.

CONTACTS AND LOCATIONS:
Overall Officials: Hira Shaukat, TDPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Cricket Board, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ripley NJ, Cuthbert M, Comfort P, McMahon JJ. Effect of additional Nordic hamstring exercise or sprint training on the modifiable risk factors of hamstring strain injuries and performance. PLoS One. 2023 Mar 2;18(3):e0281966. doi: 10.1371/journal.pone.0281966. eCollection 2023. PMID 36862645
- [Background] Maniar N, Carmichael DS, Hickey JT, Timmins RG, San Jose AJ, Dickson J, Opar D. Incidence and prevalence of hamstring injuries in field-based team sports: a systematic review and meta-analysis of 5952 injuries from over 7 million exposure hours. Br J Sports Med. 2023 Jan;57(2):109-116. doi: 10.1136/bjsports-2021-104936. Epub 2022 Dec 1. PMID 36455927
- [Background] Buchheit M, Cholley Y, Nagel M, Poulos N. The Effect of Body Mass on Eccentric Knee-Flexor Strength Assessed With an Instrumented Nordic Hamstring Device (Nordbord) in Football Players. Int J Sports Physiol Perform. 2016 Sep;11(6):721-726. doi: 10.1123/ijspp.2015-0513. Epub 2016 Aug 24. PMID 26638728
- [Background] Sugiura Y, Saito T, Sakuraba K, Sakuma K, Suzuki E. Strength deficits identified with concentric action of the hip extensors and eccentric action of the hamstrings predispose to hamstring injury in elite sprinters. J Orthop Sports Phys Ther. 2008 Aug;38(8):457-64. doi: 10.2519/jospt.2008.2575. Epub 2008 Aug 1. PMID 18678956
- [Background] Bourne MN, Duhig SJ, Timmins RG, Williams MD, Opar DA, Al Najjar A, Kerr GK, Shield AJ. Impact of the Nordic hamstring and hip extension exercises on hamstring architecture and morphology: implications for injury prevention. Br J Sports Med. 2017 Mar;51(5):469-477. doi: 10.1136/bjsports-2016-096130. Epub 2016 Sep 22. PMID 27660368
- [Background] Augustsson J, Andersson H. Differences in Peak Knee Flexor Force between Eccentric-Only and Combined Eccentric-Concentric Nordic Hamstring Exercise. Sports (Basel). 2023 Feb 7;11(2):41. doi: 10.3390/sports11020041. PMID 36828326
- [Background] Lodge C, Tobin D, O'Rourke B, Thorborg K. Reliability and Validity of a New Eccentric Hamstring Strength Measurement Device. Arch Rehabil Res Clin Transl. 2019 Nov 22;2(1):100034. doi: 10.1016/j.arrct.2019.100034. eCollection 2020 Mar. PMID 33543063